CLINICAL TRIAL: NCT03370211
Title: Effect of Resistance Training on Body Composition, Functional Capacity, Inflammatory and Oxidative Stress Biomarkers in Sarcopenic Obesity Elderly Women: a Randomized Controlled Trial
Brief Title: Resistance Training and Sarcopenic Obesity Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Crisieli Maria Tomeleri, Doctor, Universidade Estadual de Londrina
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UELGEP2017
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Sarcopenic Obesity; Inflammation; Functional Capacity
Keywords: resistance training; inflammatory markers; functional capacity
MeSH Terms: conditions — Inflammation | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental intervention (Experimental): The training group performed the resistance training (RT) program. All participants were personally supervised by physical education professionals with substantial RT experience. The sessions were performed 3 times per week on Mondays, Wednesdays, and Fridays, wirh 3 sets of 10-15 repetition maximums (RM).The RT program was performed in the following order: chest press, seated row, triceps pushdown, preacher curl, horizontal leg press, knee extension, leg curl, , and seated calf raise. Participants were afforded a 1 to 2 min rest interval between sets and 2 to 3 min between each exercise. The training load was consistent with the prescribed number of repetitions for the three sets of each exercise.
  Interventions: Other: resistance training
- control group (No Intervention): The control group did not perform any type of physical exercise during the intervention period.

INTERVENTIONS:
Other: resistance training — Participants from TG performed program, executed in 3 sets of 10-15RM, 3 times per week on Mondays, Wednesdays, and Fridays. The RT program was composed of 8 exercises comprising one exercise with free weights and seven with machines performed in the following order: chest press, horizontal leg press, seated row, knee extension, preacher curl (free weights), leg curl, triceps pushdown, and seated calf raise. All participants were personally supervised by physical education professionals with substantial RT experience to help ensure consistent and safe exercise performance. Participants were instructed to inhale during the eccentric phase and exhale during the concentric phase while maintaining a constant velocity of movement at a ratio of approximately 1:2 seconds (concentric and eccentric phases, respectively). Participants were afforded 1 to 2 min of rest between sets and 2 to 3 min between each exercise. The average duration of each session lasted approximately 50-60 minutes.
  Arms: experimental intervention

SUMMARY:
In this manuscript, we investigated the effect of resistance training (RT) on body composition, functional capacity, inflammatory and oxidative stress biomarkers in sarcopenic obesity elderly women, using a randomized controlled trial.

DETAILED DESCRIPTION:
To investigate the effects of resistance training (RT) program on body composition, functional capacity, inflammatory and oxidative stress biomarkers in sarcopenic obesity elderly women. This study is a randomized controlled trial. Thirty-seven sarcopenic obesity (SO) elderly women were randomly allocated into two groups: a training group (TG, n=18) or a non-exercising control group (CG, n=19). A supervised RT program was performed by TG for 12 weeks and CG did not perform any type of physical exercise during this period. Body composition (DXA), functional capacity [(muscular strength, and the 10 m walk test (10MW), and rising from sitting position test (RSP)] and blood sample measurements (after a 12 h fasting) were performed pre- and post-training. The investigation was carried out over a period of 16 weeks, with 12 weeks dedicated to the RT program and 4 weeks allocated for measurements. Anthropometric, muscular strength, body composition, and blood samples measurements were performed at weeks 1-2, and 15-16. A supervised progressive RT was performed between weeks 3-14. The CG did not perform any type of physical exercise during this period. However, given the possible positive effects of exercise, elderly women of this group were incorporated into a new exercise program after the end of this experiment. Data distribution was tested using the Shapiro Wilk test. Descriptive statistics are presented as means and standard deviations. Student's independent t-test and chi-square test were used to compare the control and intervention groups regarding the general characteristics and clinical conditions (categorical variables), respectively. Two-way analysis of covariance (ANCOVA) for repeated measures was applied for comparisons, with baseline scores used as covariates. When F-ratio was significant, Bonferroni's post hoc test was employed to identify the mean differences. Between group effect size (ES) was calculated to verify magnitude of the difference between groups. The Z-score of the percentage changes (from pre- to post-training) of the raw data for each parameter was calculated, and a total Z-score, derived from the all components was calculated. To verify the differences among groups on total Z-scores, a test T independent also was applied. For all statistical analyses, significance was accepted at P< 0.05. The data were analyzed using STATISTICA software version 13.2 (Statsoft Inc., Tulsa, OK, USA).

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more;
* presented sarcopenic obesity SO [which was defined by the simultaneous presence of sarcopenia and obesity (Batsis et al., 2015; Studenski et al., 2014), whereas women were considered sarcopenic if appendicular lean soft tissue (LST) <15.02 kg, and obese if percentage of body fat ≥ 35% (Batsis et al., 2015)];
* physically independent;
* free from cardiac or orthopedic dysfunction;
* not receiving hormonal replacement and/or thyroid therapy;
* not using equipment that would compromise the accomplishment of protocols and tests;
* not performing any regular physical exercise more than once a week over the six months preceding the beginning of the investigation.

Exclusion Criteria:

* individuals with any metallic implant or artificial pacemaker, who had undergone surgery, who were unable to perform the tests and trainings;
* volunteers who failed the medical examination for any reason;
* refused or were unable to give consent.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in body composition | baseline and 12 weeks
  To assess total and appendicular lean soft-tissue (LST), and total body fat (in kg), whole-body dual-energy X-ray absorptiometry DXA (Lunar Prodigy, model NRL 41990, GE Lunar, Madison, WI) was used.
Change in muscular strength | baseline and 12 weeks
  Functional capacity was evaluated using measures of muscular strength (total strength) by 1RM test assessed in the chest press (CP), knee extension (KE), and preacher curl (PC) exercises, performed in this exact order.The 1RM was recorded as the final load lifted in which the subject was able to complete only one single maximal execution. Total strength was determined by the sum of the 3 exercises and express in Kg.
Change in inflammatory biomarkers | baseline and 12 weeks
  Measurements of tumor necrosis factor alpha (TNF-α), and Interluekin-6 (IL-6), were determined by enzyme-linked immunosorbent assay (ELISA), according to the specifications of the manufacturer (Quantikine High Sensitivity Kit, R&D Systems, Minneapolis, MN) and performed in a microplate reader Perkin Elmer, model EnSpire (Waltham, MA, USA). The results are presented in picograms per milliliter (pg/ml). All samples were determined in duplicate to guarantee the precision of the results.
Change in oxidative stress biomarkers | baseline and 12 weeks
  For the oxidative stress measurements, advanced oxidation protein products (AOPP) were determined in the plasma using a semiautomatic method described by Witko-Sarsat et al. (Witko-Sarsat et al., 1996). AOPP concentrations are expressed as micromoles per liter (μmol/L) of chloramines-T equivalents.
Change in functional capacity | baseline and 12 weeks
  Functional capacity was evaluated using measures of muscular strength (total strength), the 10-m walk test (10MW) and rising from sitting position test (RSP) express in (s). For the 10MW test older women were required to walk the distance of 10 m rapidly to evaluate the displacement speed; for the RSP, they were required to get up and sit down from a chair five times consecutively. In both tests the timer was triggered after the command "start now". At the moment the task was completed the timer was stopped.
Change in insulin-like growth factor 1 (IGF-1) | baseline and 12 weeks
  The concentrations of insulin-like growth factor 1 (IGF-1), were obtained in a specialized laboratory by a chemiluminescence method using a Liaison XL Immunoassay Analyzer (DiaSorin S.p.A, Saluggia, Italy). The values are expressed in (µU/mL)

SECONDARY OUTCOMES:
Change in C-reative protein (CRP) | baseline and 12 weeks
  Measurements of serum levels of high-sensitivity CRP were carried out using a biochemical auto-analyzer system (Dimension RxL Max - Siemens Dade Behring) according to established methods in the literature consistent with the manufacturer's recommendations. The results are presented in milligram/liter (mg/L)
Changes in Anthropometry Parameters | baseline and 12 weeks
  Body mass was measured to the nearest 0.1 kg using a calibrated electronic scale (Balmak, Laboratory Equipment Labstore, Curitiba, Paraná, Brazil), with the participants wearing light workout clothing and no shoes. Height was measured with a stadiometer attached to the scale to the nearest 0.1 cm, with subjects standing without shoes. Body mass index was calculated as body mass in kilograms divided by the square of height in meters.

IPD SHARING:
Plan to Share IPD: No